CLINICAL TRIAL: NCT05098431
Title: Comparison of Three Approaches of Motor Evoked Potential Recording to Detect a More Reliable Measure to Predict and Prevent Nerve Damage During Spine Surgery
Brief Title: Comparison of Three Approaches of Electrode Placement to Detect Changes in Motor Evoked Potentials During Spine Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll patients.
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1565509
Record Dates: First submitted 2021-09-09; First posted 2021-10-28 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Stenosis; Spinal Curvatures; Spondylitis; Spondylosis
Keywords: Intraoperative Neuromonitoring; Motor Evoked Potential
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Spinal Stenosis; Spinal Curvatures; Spondylitis; Spondylosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental Arm (Experimental): Receive Quadriceps MEPs during procedure
  Interventions: Other: Quadriceps and Rectus Femoris MEP Recording

INTERVENTIONS:
Other: Quadriceps and Rectus Femoris MEP Recording — Participants will receive additional electrodes placed intramuscularly to facilitate three separate approaches of quadriceps MEP recording

SUMMARY:
Motor Evoked Potentials are an aspect of intraoperative neuromonitoring, a tool used by neurophysiologists during surgery to prevent irreversible damage to the spinal cord during procedures. This study investigates the utility of three separate quadriceps MEP recording approaches over a total of 40 limbs (20 participants).

DETAILED DESCRIPTION:
The long-term objective of this research is to understand how differing recording techniques may enhance the ability to accurately identify clinically relevant changes in Motor Evoked Potentials (MEPs) during a variety of surgeries where the central motor tracts or lumbar spinal roots are at risk.The specific aims of the proposed research are:

1. Using transcranial magnetic stimulation, evaluate the effects on compound muscle action potentials utilizing intramuscular bipolar recording vs subdermal referential recordings vs subdermal bipolar recordings.
2. Evaluated the variability of amplitude and area between the intramuscular and subdermal recording techniques.

The initial focus will be on recording techniques to obtain stable MEPs in a proximal lower limb muscle, specifically the quadriceps. Continuation research may focus on stimulation techniques to facilitate proximal MEPs and ultimately to improved specificity of MEP changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years of age
* Patients must be undergoing thoracic or lumbar spine surgery where quadriceps MEP recording would be the standard of care
* Patients should have normal preoperative quadriceps strength
* Patients are capable of understanding the informed consent and have signed the informed consent document prior to any study-specific screening procedures or evaluations being performed

Exclusion Criteria:

* Patients with ongoing psychiatric concerns would be excluded.
* Patients who are non-English speakers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Motor Evoked Potentials recorded with an Intramuscular bipolar electrodes in the Rectus Femoris | Duration of surgery
  MEPs will be evoked throughout the duration of the surgery. MEPs will be recorded in the Rectus Femoris using intramuscular bipolar electrodes.
Motor Evoked Potentials recorded with a subcutaneous referential electrodes in the Rectus Femoris | Duration of surgery
  MEPs will be evoked throughout the duration of the surgery. Electrodes will be placed in the Rectus Femoris to serve as a reference.
Motor Evoked Potentials recorded with secondary subcutaneous referential electrodes in the Rectus Femoris | Duration of surgery
  MEPs will be evoked throughout the duration of the surgery. Electrodes will be placed in the Rectus Femoris to serve as a reference.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Strommen, MD, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No